CLINICAL TRIAL: NCT00218595
Title: Evaluation of Dialectical Behavior Therapy in Treatment of Opioid Addiction and Emotional Problems
Brief Title: DBT Compared to I/GDC for the Treatment of Opiate Addiction in Emotionally Dysregulated Patients. - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00010957; 5R01DA026454-03 (NIH); R01-17372-1
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2013-01

CONDITIONS: Dialectical Behavior Therapy; Individual and Group Drug Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DBT (Experimental)
  Interventions: Behavioral: DBT
- I/GDC (Active Comparator)
  Interventions: Behavioral: I/GDC

INTERVENTIONS:
Behavioral: DBT — Dialectical behavior therapy plus opiate replacement medication.
  Arms: DBT
Behavioral: I/GDC — Individual and group drug counseling plus opiate replacement medication.
  Arms: I/GDC

SUMMARY:
The purpose of this study is to examine the efficacy of DBT compared to a standard drug counseling approach for the treatment of opiate addiction and borderline personality disorder (BPD). Treatment research has repeatedly shown that retention of BPD and substance addicted individuals to be the among the most challenging for therapists. DBT has established itself as one of the most effective treatments for treatment retention of these patients and for reducing parasuicidal and self-injurious behaviors.

This study is one of two in a multi-site RCT for the treatment of opiate addiction. DBT has been shown to be efficacious for the treatment of BPD patients and it has been extended in this study to target addictive behaviors in these patients. The study consists of three treatment parts: weekly individual and group therapy and suboxone maintenance medication. Participants are provided therapy on a weekly basis for one year and suboxone for 2 years. Assessments for tracking outcome are conducted every 4 months.

It is hypothesized patients in the DBT condition will show a reduction of substance use, parasuicidal and other psychological difficulties and these gains will be maintained through the year of follow-up assessments. In addition, it is predicted that adherence to DBT treatment protocols will be associated with improved outcomes. Finally, it is predicted that treatment "dosage" (average hours of therapy/week) will be positively related to clinical improvement.

DETAILED DESCRIPTION:
The study design is a two arm randomized clinical trial comparing a one year treatment program of Dialectical Behavior Therapy (DBT) + suboxone for heroin addicted individuals meeting criteria for borderline personality disorder (BPD) to a one year program of standard drug counseling (I/GDC) + suboxone. Drug counseling will consist of manualized individual sessions + group therapy. Participants in both conditions will be prescribed psychotropic medications following a standardized medication protocol developed specifically for BPD individuals. Each site will enroll 86 clients with both treatment conditions being conducted at each site. Assessments measuring drug use, suicidal behaviors, retention and other treatment-related behaviors, general psychopathology and functioning, and increases in behavioral skills will be given at four month intervals for two years

There are five outcome domains of principal interest in this study:

1. Drug use: The primary outcome measure here is proportions of urinalysis (UA) coded positive for opiates;
2. Suicidal behaviors: The primary outcome measure here is number of suicides + suicide attempts. The domain of suicidal behaviors also includes (a) the number, medical risk, risk/rescue score and suicide intent of all parasuicide, (b) the number of suicide threats and suicide crises, and (c) the level of suicidal ideation and suicide intent;
3. Therapy-interfering behaviors: The primary outcome measure here is maintenance in therapy;
4. Quality of life interfering behaviors: The primary outcome measure here is combined number of days on a psychiatric inpatient unit + days in jail (THI, SHI);
5. Behavioral skills: The primary outcome measure here is the DBT Skills scale score from the Revised Ways of Coping Checklist (RWCCL);
6. Risky sexual behavior: the primary outcome measure here is the number of risky sexual behaviors in the time period [Casual Partners questionnaire revised [CPQ-R] and diary card].

ELIGIBILITY:
Inclusion Criteria:

1. Meets SCID-I criteria for opiate dependence.
2. Meets IPDE and SCID criteria for BPD (DSM-IV)
3. Over 18 years old
4. Resides within commuting distance of treatment
5. Consents to outpatient treatment for drug addiction

Exclusion Criteria:

1. Bipolar, Schizophrenia, Schizophreniform, or Schizoaffective Disorders, Psychosis NOS
2. IQ less than 70; life threatening anorexia; current and chronic absence of shelter; impending jail/prison for more than three weeks (problems which by their presence or severity preclude ability to attend or understand treatment and/or requires priority treatment over SUD treatment)
3. Court order to treatment, court order to treatment or to jail, or agency order to treatment or loss of child custody (due to consequent inability to freely drop-out of treatment)
4. Is pregnant, plans to become pregnant during treatment phase, or becomes pregnant before random assignment to study condition
5. Is unable to tolerate suboxone induction phase
6. Is currently stable on an adequate dose of methadone
7. Current benzodiazepine abuse or dependence
8. Refuses: to discontinue current mental health or drug abuse treatment or random assignment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Psychological assessment interview | Baseline, 4-month, 8-month, 12-month, 16-month, 20-month, 24-month
Urinalysis | 3x/week during active treatment; 1x/week during follow-up year

SECONDARY OUTCOMES:
Pre- and post-session therapist and client questionnaires | 1x/week during active treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Rosenthal, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States